CLINICAL TRIAL: NCT04007276
Title: The Effect of Lumify™ (Brimonidine Tartrate Ophthalmic Solution 0.025%) on Ocular Redness, Intraocular Pressure, and Eyelid Position in Glaucoma Patients Using Brimonidine 0.2%, 0.15%, or 0.1%
Brief Title: The Effect of Lumify™ on Ocular Redness, Intraocular Pressure, and Eyelid Position in Glaucoma Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tulane University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Lumify Study
Record Dates: First submitted 2019-06-26; First posted 2019-07-05 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Glaucoma; Glaucoma, Open-Angle; Glaucoma; Drugs; Droopy Eyelid; Ptosis; Glaucoma, Primary Open Angle
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Blepharoptosis | interventions — Brimonidine Tartrate

STUDY DESIGN:
Intervention Model Description: Each patient will be randomized to receive the study medication in one eye and placebo in the other eye.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lumify Arm (Experimental): In each subject, each eye will be randomized to receive a single drop of either Lumify™ (brimonidine tartrate ophthalmic solution 0.025%) or a sterile balanced saline solution.
  Interventions: Drug: brimonidine tartrate ophthalmic solution 0.025%
- Control Arm (Sham Comparator): In each subject, each eye will be randomized to receive a single drop of either Lumify™ (brimonidine tartrate ophthalmic solution 0.025%) or a sterile balanced saline solution.
  Interventions: Other: sterile balanced saline solution

INTERVENTIONS:
Drug: brimonidine tartrate ophthalmic solution 0.025% — Single dose of brimonidine tartrate ophthalmic solution 0.025% applied as an eye drop to the eye surface.
  Other Names: Lumify™
  Arms: Lumify Arm
Other: sterile balanced saline solution — Single dose of sterile balanced saline solution applied as an eye drop to the eye surface.
  Arms: Control Arm

SUMMARY:
Glaucoma represents a group of conditions that cause damage to the optic nerve and can lead to irreversible vision loss. Current treatments are aimed at lowering intraocular pressure while minimizing medication side effects. Lumify™ (Brimonidine Tartrate Ophthalmic Solution 0.025%) is an FDA-approved medication for alleviating eye redness, a common side effect of glaucoma medications. The purpose of this study is to evaluate the effect of Lumify™ on eye redness, intraocular pressure, and eyelid position in patients with glaucoma who are already using the Brimonidine 0.1%, 0.15% or 0.2% eye drops.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis of primary open angle glaucoma
* Willing and able to give informed consent
* Current and greater than 6 weeks of brimonidine 0.2%, 0.15% or 0.1% use

Exclusion Criteria:

* Pregnancy
* Prisoners
* Known allergy or sensitivities to brimonidine
* No surgery within the past 6 months
* No history of lid surgery or botox
* Any other significant ophthalmologic disorder or condition with relevant effect on ocular redness, IOP, or eyelid position as evaluated by principal investigator
* Inability to sit comfortably for 30 minutes
* Prior use of eye whiteners (eg, vasoconstrictors), decongestants, antihistamines, or phenylephrine dilating drops within 1 week of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-11-10 (Estimated); Primary Completion 2031-06-01 (Estimated); Study Completion 2036-06-01 (Estimated)

PRIMARY OUTCOMES:
Ocular redness | 5 minutes after application of eye drop
  Scoring of ocular redness on clinical photographs using the the Investigator Ocular Redness Scale (0-4; 0 = no ocular redness, 4 = extremely severe ocular redness)
Ocular redness | 15 minutes after application of eye drop
  Scoring of ocular redness on clinical photographs using the the Investigator Ocular Redness Scale (0-4; 0 = no ocular redness, 4 = extremely severe ocular redness)
Ocular redness | 30 minutes after application of eye drop
  Scoring of ocular redness on clinical photographs using the the Investigator Ocular Redness Scale (0-4; 0 = no ocular redness, 4 = extremely severe ocular redness)
Ocular redness | 60 minutes after application of eye drop
  Scoring of ocular redness on clinical photographs using the the Investigator Ocular Redness Scale (0-4; 0 = no ocular redness, 4 = extremely severe ocular redness)
Intraocular pressure | 60 minutes after application of eye drop
  Measurement of intraocular pressure using handheld tonometer (TonoPen)

SECONDARY OUTCOMES:
Palpebral fissure height | 60 minutes after application of eye drop
  Measurement of distance between inner margin of upper and lower eyelids from clinical photographs
Eye discomfort | 60 minutes after application of eye drop
  Subjective scoring of ocular discomfort by patient on a 0-10 unit scale (0 = very comfortable, 10 = very uncomfortable)

CONTACTS AND LOCATIONS:
Overall Officials: Ze Zhang, MD, Principal Investigator — Tulane University
Locations (1):
- Tulane University Medical Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No